CLINICAL TRIAL: NCT04893304
Title: Study of the Effect of Fractional co2 Laser Versus Q Switched:NdYAG Laser in the Treatment of Acanthosis Nigricans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Fahim, Principale investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAS123
Record Dates: First submitted 2021-04-25; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Acanthosis Nigricans
MeSH Terms: conditions — Acanthosis Nigricans | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 group of 20 patients doing both types of lasers on 2 sites (Other): comparing both types of laser
  Interventions: Device: co2 laser

INTERVENTIONS:
Device: co2 laser — types of laser
  Other Names: NdYAG laser

SUMMARY:
This prospective randomized comparative split study will be conducted at the outpatient clinic, Dermatology department, Faculty of Medicine, Cairo University and will include 20 patients with acanthosis nigricans in otherwise healthy individuals which will be recruited and assessed for eligibility for inclusion according to the above criteria.

-Evaluation:

All patients will be subjected to:

Pre-operative preparation:

* Informed written consent will be taken from every patient prior to the study.
* Detailed history taking including onset, course, duration of the disease and occupation (sun-exposed or not), predisposing factors, history of keloid tendency, associated diseases and previous treatments.
* Assessment of skin type, BMI, degree of AN, HbA1C, site of lesions in all patients and degree of improvement.
* Photography: will evaluate the clinical response to treatment for each patient Photos will be taken before starting the study, before every session, and two weeks after the last session.
* Melanin index (MI) will be measured using reflectance spectrophotometer in order to assess the degree of hyperpigmentation before starting the study and two weeks after the last session. Research Template 8 Final Version: April 2019
* Acanthosis Nigricans Area and Severity Index (ANASI) score (Zaki et al., 2018) will be done for all patients before starting the study and two weeks after the last session.
* Patient satisfaction score will be assessed before starting the study and two weeks after the last session.
* Patient evaluation (clinical percentage of improvement).

Operation :

One side of the affected area will be randomly assigned to fractional CO2 laser every four weeks for three months. The other side will be assigned to Q-switched Nd:YAG laser every four weeks for three months.

Method of randomization:

Using closed envelopes containing cards with fractional CO2 Rt and fractional CO2 Lt and the patient will draw one of them blindly. The assessment will be done by blinded investigator. Post-operative: Patients will be instructed to avoid sun exposure for one week after the session and regular use of sun block in between sessions.

DETAILED DESCRIPTION:
This prospective randomized comparative split study will be conducted at the outpatient clinic, Dermatology department, Faculty of Medicine, Cairo University and will include 20 patients with acanthosis nigricans in otherwise healthy individuals which will be recruited and assessed for eligibility for inclusion according to the above criteria. -Evaluation:

All patients will be subjected to the following:

Pre-operative preparation:

Informed written consent will be taken from every patient prior to the study. Detailed history taking including onset, course, duration of the disease and occupation (sun-exposed or not), predisposing factors, history of keloid tendency, associated diseases and previous treatments.

Assessment of skin type, BMI, degree of AN, HbA1C, site of lesions in all patients and degree of improvement.

Photography: will evaluate the clinical response to treatment for each patient Photos will be taken before starting the study, before every session, and two weeks after the last session.

Melanin index (MI) will be measured using reflectance spectrophotometer in order to assess the degree of hyperpigmentation before starting the study and two weeks after the last session. Research Template 8 Final Version: April 2019 Acanthosis Nigricans Area and Severity Index (ANASI) score (Zaki et al., 2018) will be done for all patients before starting the study and two weeks after the last session.

Patient satisfaction score will be assessed before starting the study and two weeks after the last session.

Patient evaluation (clinical percentage of improvement).

Operation :

One side of the affected area will be randomly assigned to fractional CO2 laser every four weeks for three months. The other side will be assigned to Q-switched Nd:YAG laser every four weeks for three months.

Method of randomization:

Using closed envelopes containing cards with fractional CO2 Rt and fractional CO2 Lt and the patient will draw one of them blindly. The assessment will be done by blinded investigator.

Post-operative: Patients will be instructed to avoid sun exposure for one week after the session and regular use of sun block in between sessions.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 18 years old
2. both genders
3. skin type III to V
4. controlled diabetus

Exclusion Criteria:

1. pregnancy and lactation
2. scarring
3. active skin infections
4. endocrinal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
patient evaluation | 3 months
  Acanthosis nigricans area and severity index is scoring system used to assess patients before the session and after the session to assess finally the improvement

IPD SHARING:
Plan to Share IPD: Yes
results and discussion can be shared
Time Frame: after finishing the paper and will be always be available
Access Criteria: through the pubmed